CLINICAL TRIAL: NCT02263742
Title: Increasing Health Care Choices and Improving Health Outcomes Among Persons With Serious Mental Illness
Brief Title: Project Wellness Enhancement: Increasing Health Care Choice and Outcomes for People With Mental Illness
Acronym: WE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1310012851
Record Dates: First submitted 2014-03-31; First posted 2014-10-13 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Mental Health Wellness 1; Mental Illnesses; Other Diagnoses, Comorbidities, and Complications | Patient
Keywords: Healthcare choice and outcomes; Peer-led whole health; Mental Illness; Peer Health Navigation; Health care Coordination
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer whole health (Experimental): Peer whole health intervention will be compared to the treatment as usual at Wellness Center to assess healthcare choice and outcomes
  Interventions: Behavioral: Peer whole health intervention
- EBPs at Wellness Center (Active Comparator): EBPs at Wellness Center will be the active comparative to measure healthcare choice and outcomes with the peer whole health intervention
  Interventions: Behavioral: EBPs at Wellness Center

INTERVENTIONS:
Behavioral: Peer whole health intervention — Provide wraparound peer support, education, and navigation to individuals
  Arms: Peer whole health
Behavioral: EBPs at Wellness Center — four EBPs: a) on-site primary care; b) screening of clients for modifiable risk factors and medical conditions; c) care coordination; and d) peer health navigation
  Arms: EBPs at Wellness Center

SUMMARY:
This project aims to study health outcomes of individuals with mental illness attending a co-located primary health care center in a mental health center. This study uses mixed methods to collect a range of information about who chooses to use what Wellness Center services and in what combinations, with what short and longer-term effects and with what outcomes.

Based on participant interviews, identify barriers to and facilitators of access, service, and improvements in person-centered outcomes and elicit suggestions for enhancing health care outcomes and choice.

Collaborate with persons in recovery in using the data collected through Aims 1 and 2 to develop and pilot the effectiveness of a new peer-led community based intervention in enhancing access and choice and improving person-centered health outcomes.

DETAILED DESCRIPTION:
Background: Americans with serious mental illnesses (SMI) die an average of 25 years earlier due to modifiable risk factors, medical conditions, and lack of access to quality, coordinated care. Strategies for addressing this disparity have amassed evidence. What remains to be determined is who will choose to use these evidence-based practices (EBPs) when implemented in routine practice, in what combinations, with what short term effects and health outcomes, and what else might be needed for persons for whom these strategies are not effective.

Objectives: The proposed research builds upon the investigators receipt of a SAMHSA grant that established an integrated Wellness Center (WC) within the local mental health center that provides four EBPs: a) on-site primary care; b) screening of clients for modifiable risk factors and medical conditions; c) care coordination; and d) peer health navigation. Through PCORI, the investigators propose to add a comparative effectiveness dimension and a focus on patient-centered outcomes. The investigators specific aims are:

1. to assess patient preferences and use of services, short-term effects, and longer term outcomes associated with various practices for the population and subpopulations;
2. to identify barriers to and facilitators of access, service use, and improvements in traditional and patient-centered health outcomes; and
3. to develop and pilot a peer-led, community-based intervention in enhancing access and choice, and improving patient-centered health outcomes, among 40 treatment-refractory clients of the WC.

The investigators long-term objectives are to: a) identify which practices work for which persons with SMI in improving health and patient-centered outcomes, and b) provide stakeholders around the nation with the knowledge and tools to replicate this model efficiently, effectively, and broadly.

Methods: The sample includes 360 poor, urban adults with SMI who are at risk for or have co-morbid medical conditions. Using participatory and mixed methodology, the investigators will assess Specific Aims 1 & 2 by collecting health and patient-centered outcome data on patients entering the WC and at 6 month follow-up intervals and analyze the data using Linear Mixed Models and logistic regression. Outcome data from the pilot intervention (Aim 3; N=40) will be compared to outcomes of a propensity matched sample of WC patients. Qualitative data will be collected each year through focus groups (N=48 agency stakeholders, year 1) and individual interviews (50 WC patients, years 2 & 3).

Projected Patient Outcomes: Outcomes include both traditional medical/clinical outcomes (e.g., blood pressure, BMI, fasting plasma glucose, HbGA1c, cholesterol, triglycerides, alcohol and drug use, psychiatric symptoms) and a range of patient-centered outcomes to be identified by key stakeholders in the initial phase of research. The investigators previous research suggests that these outcomes are likely to include self-efficacy, quality of life, employment, citizenship, and social connectedness.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Clients receiving services from CMHC and the Wellness Center.
* Research staff will verify with CMHC staff that the potential participant is receiving services currently at CMHC.
* Provider research subjects will be included if they are a mental health provider at CMHC or if they are members of the staff for the Wellness Center
* Adults with serious mental illness and physical illness

Exclusion Criteria:

* Participant research subjects not receiving services at CMHC and the Wellness Center
* Provider research subjects of other agencies will be excluded
* Children and youth under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Effectiveness of a Co-located Primary Health Care Center in a Local mental health center | up to 30 months
  Use mixed methods to collect a rage of information about who chooses to use Using quantitative and qualitative measures by looking at the number of participants, follow up rates, improvement in health indices

SECONDARY OUTCOMES:
Effectiveness of health care navigation in improving health outcomes for people with mental illness | up to 30 months
  Use mixed methods to collect a rage of information about who chooses to use Using quantitative and qualitative measures by looking at the number of participants, follow up rates, improvement in health indices, including some patient centered measures, and also the number of times they meet with their health care navigators
Universal Health screening | up to 30 months
  Look at whether clients of the Wellness Center have improvement in their overall health by looking at their health measurements and lab works from each of their 6 month appointments

OTHER OUTCOMES:
Collaborate with persons in recovery in using data collected to develop and pilot a new peer led, community based intervention in enhancing access and choice | up to 30 months
  48 participants will be in a pilot intervention run by peers on whole health, measures will be both qualitative and quantitative to look for overall health improvement and choices

CONTACTS AND LOCATIONS:
Overall Officials: Chyrell Bellamy, Ph.D., Principal Investigator — Yale University; Kimberly D Antunes, BSW, Study Director — Yale University
Locations (2):
- United States (2):
  - CT Mental Health Center, New Haven, Connecticut
  - Yale University Program for Recovery and Community Health, New Haven, Connecticut